CLINICAL TRIAL: NCT06816134
Title: A Prospective, Randomized Controlled Clinical Study on the Efficacy and Safety of the TmBU Regimen Versus mBUCY Regimen for Conditioning Before Allo-HSCT in High-risk or Relapsed/Refractory Acute Leukemia
Brief Title: Study on the Efficacy and Safety of the TmBU Conditioning Regimen in High-risk or Relapsed/Refractory Acute Leukemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, Sheng-Li Xue, MD, Prof., The First Affiliated Hospital of Soochow University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SZConditioning01
Record Dates: First submitted 2025-02-04; First posted 2025-02-10 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia; Transplantation, Stem Cell; Conditioning Therapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Control Groups

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TmBu conditioning Regimen Group (Experimental): TmBU conditioning regimen（TT 9mg/kg -8~-7d; Ara-C 2g/m2/d -6d; CDA 5 mg/m2/d -6d; Bu 3.2 mg/kg/d from -5 to -3 days）
  Interventions: Drug: TmBU conditioning Regimen
- mBUCY conditioning Regimen Group (Active Comparator): mBuCy conditioning regimen（CCNU/BCNU -9d, Ara-C 2g/m2/d -8d; CDA 5 mg/m2/d -8d; Busulfan 3.2 mg/kg/d from -7 to -5 days; Cyclophosphamide 1.8 mg/m2/d from -4 to -3 days）
  Interventions: Drug: mBUCY conditioning regimen

INTERVENTIONS:
Drug: TmBU conditioning Regimen — TmBU conditioning Regimen and GVHD Prophylaxis of Haploid transplantation (Haplo-HSCT) and unrelated donor transplantation (UDT) : Cyclosporine A (CsA) + Mycophenolate mofetil dispersible tablets (MMF) + short-term low-dose methotrexate (MTX) + rabbit anti-human antithymocyte globulin (ATG) or GVHD Prophylaxis of Matched Sibling Donor Hematopoietic Stem Cell Transplantation (MSD-HSCT)：Cyclosporine A (CsA) + short-term low-dose methotrexate (MTX), then stem cells are infused into patient's blood.
  Other Names: Experimental Group
  Arms: TmBu conditioning Regimen Group
Drug: mBUCY conditioning regimen — mBUCY conditioning Regimen and GVHD Prophylaxis of Haploid transplantation (Haplo-HSCT) and unrelated donor transplantation (UDT): Cyclosporine A (CsA) + Mycophenolate mofetil dispersible tablets (MMF) + short-term low-dose methotrexate (MTX) + rabbit anti-human antithymocyte globulin (ATG) or GVHD Prophylaxis of Matched Sibling Donor Hematopoietic Stem Cell Transplantation (MSD-HSCT)：Cyclosporine A (CsA) + short-term low-dose methotrexate (MTX), then stem cells are infused into patient's blood.
  Other Names: Control Group
  Arms: mBUCY conditioning Regimen Group

SUMMARY:
This project is a prospective, single-center, randomized controlled clinical study. The subjects were high-risk or relapsed/refractory AML or ALL patients aged ≤ 65 years diagnosed by bone marrow cell morphology, immunology, genetics and therapeutic efficacy evaluation. The TmBU scheme or modified Bu/Cy (mBuCy) scheme was used for pretreatment in allo-HSCT. The primary endpoint of the study was the 2-year cumulative incidence of relapse (CIR) after allo-HSCT, and the secondary endpoints were 2-year overall survival rate (OS), progressing-free survival rate (PFS), non-relapse mortality rate (NRM), graft-versus-host disease (GVHD)-free relapse-free survival (GRFS) rate.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of AML or ALL according to WHO 2022 guideline criteria, with indications for allo-HSCT list below:

  1. Relapsed/primary refractory (definitions refer to NCCN 2025) or genetic high-risk group AML at diagnosis (risk stratification refers to ELN 2022)
  2. High-risk at diagnosis (risk stratification refers to ELN 2022) or MRD positive before transplantation B-ALL
  3. Confirmed diagnosis of T-ALL
  4. History of central nervous system leukemia (CNSL) or histopathologically confirmed extramedullary manifestation (EMD) during the course of the AML or ALL
* Age 15-65 years old (≤ 65 years old)
* HCT-CI score < 2 points ECOG 0-2 points
* Adequate organ function:

  1. Cardiac NYHA grade ≤ 2, left ventricular ejection fraction ≥55%
  2. Creatinine clearance ≥ 50ml/min
  3. ALT and AST ≤ 2.5 times the upper limit of the normal range, and total bilirubin ≤ 1.5 times the upper limit of the normal range
  4. Oxygen saturation > 92% without oxygen
* Expected survival time ≥ 3 months
* Ability to understand and voluntarily sign the informed consent form

Exclusion Criteria:

* With other malignant tumors and have received any treatment for this tumor within the past 3 years
* Previous or current other CNS disease (such as epilepsy, generalized seizure disorder, paresis, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or psychosis) or any CNS-related autoimmune disease
* HIV/Syphilis infection or uncontrolled active other infections (bacteria or fungus or virus is included)
* With active hepatitis B or hepatitis C infection
* Patients received cardiac angioplasty or stent implantation within 12 months before signing the informed consent form, or have symptoms requiring medical treatment for coronary heart disease
* With primary immunodeficiency or active autoimmune disease
* Previous history of severe immediate hypersensitivity reactions to any of the drugs to be used in this study
* Received a live vaccine within 6 weeks prior to screening
* Pregnant, lactating females and patients of childbearing potential who are unwilling to use contraception
* Inability to cooperate with the requirements of study, treatment and monitoring due to psychiatric illness or other conditions
* Patients not suitable for the study according to the investigator's assessment

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2028-01-30 (Estimated); Study Completion 2030-01-30 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of relapse（CIR） | 2 years
  It is measured the date from complete remission after transplantation to hematological relapse or molecular relapse was recorded. Patients who had no relapse at the last follow-up were considered as censored data, and non-relapse death was regarded as a competing risk event.

SECONDARY OUTCOMES:
Time period for hematopoietic reconstruction | 24 weeks
  Granulogenetic hematopoietic reconstitution: The absolute neutrophil count in peripheral blood needs to reach or exceed 0.5×10^9 cells/L for 3 consecutive days. Megakaryotic hematopoietic reconstitution: platelet count needs to be more than 20×10^9/L and does not rely on platelet transfusion for 7 consecutive days.
Incidence of acute graft-versus-host disease (aGVHD) | 100 days
Progressing-free survival（PFS） | 2 years
  It is measured from the date of achievement of a remission until the date of relapse from CR, or CRi, or death from any cause; patients not known to have any of these events are censored on the date they were last examined.
Overall survival（OS） | 2 years
  It is measured from the date of entry into this trial to the date of death from any cause; patients not known to have died at last follow-up are censored on the date they were last known to be alive.
Non-relapse mortality（NRM） | 2 years
  It is described as proportion of deaths due to non-primary recurrence from enrollment start date to 2 years post-transplant.
Graft-versus-host disease (GVHD)-free relapse-free survival (GRFS) | 2 years
  It is defined as a composite end point of death from any cause, relapse of malignancy, grade 3 to 4 acute GVHD, or chronic GVHD requiring systemic immune suppression therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Sheng-Li Xue, M.D., Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China